CLINICAL TRIAL: NCT00345371
Title: Phase 2, Double-Blind, Placebo-Controlled Trial of Topiramate for the Treatment of Methamphetamine Dependence
Brief Title: Topiramate for the Treatment of Methamphetamine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-CSP-1025-1; NCT00431652 (obsolete NCT alias)
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Methamphetamine
Keywords: methamphetamine addiction
MeSH Terms: interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Topiramate (Active Comparator): Subjects will receive topiramate (in tablet form) up to 200 mg/day for 13 weeks.
  Interventions: Drug: Topiramate
- Placebo Oral Tablet (Placebo Comparator): After randomization subjects will receive topiramate matched placebo (in tablet form), up to 200 mg/day for 13 weeks.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Topiramate
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo Oral Tablet
  Arms: Placebo Oral Tablet

SUMMARY:
The purpose of this study is to assess the efficacy and safety of topiramate as compared to placebo in reducing methamphetamine use in subjects with methamphetamine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Treatment seeking individuals as the time of the study
* Must be able to proved written informed consent
* Must have a body mass index greater than 18 kg/m(2)
* Must meet DSM-IV criteria for methamphetamine dependence
* Must currently be using methamphetamine as confirmed by a positive urine test over the past 14 days
* If female of child bearing potential, must agree to use birth control

Exclusion Criteria:

* Please contact the site for more information

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-04; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, Principal Investigator — VA Medical Center
Locations (8):
- United States (8):
  - Matrix Institute on Addictions, Costa Mesa, California
  - South Bay Treatment Center, San Diego, California
  - Torrance Site, Torrance, California
  - John A. Burns School of Medicine, Honolulu, Hawaii
  - Powell Chemical Dependency Center, Des Moines, Iowa
  - University of Missouri - Kansas City, Kansas City, Missouri
  - Salt Lake City VA Medical Center, Salt Lake City, Utah
  - UVA CARE, Charlottesville, Virginia

REFERENCES:
- [Background] Elkashef A, Kahn R, Yu E, Iturriaga E, Li SH, Anderson A, Chiang N, Ait-Daoud N, Weiss D, McSherry F, Serpi T, Rawson R, Hrymoc M, Weis D, McCann M, Pham T, Stock C, Dickinson R, Campbell J, Gorodetzky C, Haning W, Carlton B, Mawhinney J, Li MD, Johnson BA. Topiramate for the treatment of methamphetamine addiction: a multi-center placebo-controlled trial. Addiction. 2012 Jul;107(7):1297-306. doi: 10.1111/j.1360-0443.2011.03771.x. Epub 2012 Feb 28. PMID 22221594
- [Derived] Li MD, Wang J, Niu T, Ma JZ, Seneviratne C, Ait-Daoud N, Saadvandi J, Morris R, Weiss D, Campbell J, Haning W, Mawhinney DJ, Weis D, McCann M, Stock C, Kahn R, Iturriaga E, Yu E, Elkashef A, Johnson BA. Transcriptome profiling and pathway analysis of genes expressed differentially in participants with or without a positive response to topiramate treatment for methamphetamine addiction. BMC Med Genomics. 2014 Dec 12;7:65. doi: 10.1186/s12920-014-0065-x. PMID 25495887
- See also: Link to abstract — https://www.ncbi.nlm.nih.gov/pubmed/22221594

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate: Subjects will receive topiramate (in tablet form) up to 200 mg/day for 13 weeks.
  Topiramate
- Placebo Oral Tablet: After randomization subjects will receive topiramate matched placebo (in tablet form), up to 200 mg/day for 13 weeks.
  Placebo Oral Tablet
Period: Overall Study
Arm/Group | Topiramate | Placebo Oral Tablet
Started | 69 | 71
Completed | 39 | 38
Not Completed | 30 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo Oral Tablet | Total
Number analyzed (Participants) | 69 | 71 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (8.83) | 37.5 (8.47) | 38 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 41 | 48 | 89
Region of Enrollment [Number; unit: participants]
  United States | 69 | 71 | 140

OUTCOME MEASURES:

1. Primary Outcome: Abstinence (Weeks 6 - 12)
Description: The number of participants who abstained from methamphetamine from weeks 6 through 12
Time Frame: weeks 6 through 12
Measure: Count of Participants; unit: Participants
Arm/Group | Topiramate | Placebo Oral Tablet
Number analyzed (Participants) | 69 | 71
Participants
  Week 6 | 49 | 49
  Week 7 | 43 | 48
  Week 8 | 46 | 45
  Week 9 | 40 | 41
  Week 10 | 38 | 33
  Week 11 | 36 | 38
  Week 12 | 34 | 32

2. Secondary Outcome: Abstinence (Weeks 1 - 12)
Description: Number of participants who abstained from methamphetamine from weeks 1 through 12
Time Frame: Weeks 1 through 12
Measure: Count of Participants; unit: Participants
Arm/Group | Topiramate | Placebo Oral Tablet
Number analyzed (Participants) | 69 | 71
Participants
  Week 1 | 58 | 53
  Week 2 | 56 | 50
  Week 3 | 55 | 50
  Week 4 | 55 | 50
  Week 5 | 56 | 51
  Week 6 | 49 | 49
  Week 7 | 43 | 48
  Week 8 | 46 | 45
  Week 9 | 40 | 41
  Week 10 | 38 | 33
  Week 11 | 36 | 38
  Week 12 | 34 | 32

ADVERSE EVENTS:
Arm/Group | Topiramate | Placebo Oral Tablet
Serious Adverse Events (participants affected / at risk) | 3/69 | 8/71
Other Adverse Events (participants affected / at risk) | 63/69 | 64/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=69) | Placebo Oral Tablet (N=71)
Superficial Cutting (Psychiatric disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0)
Infected Boil (Infections and infestations) | 1 (1) | 0 (0)
Malignant hypertention (with angina) (Cardiac disorders) | 0 (0) | 1 (1)
Visual Disturbance (Eye disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Assault (Social circumstances) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abnormal ECG (Cardiac disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=69) | Placebo Oral Tablet (N=71)
Headache (Nervous system disorders) | 33 (76) | 30 (68)
Fatigue (General disorders) | 20 (22) | 14 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 11 (14)
Diarrhea (Gastrointestinal disorders) | 11 (14) | 8 (12)
Dizziness (Nervous system disorders) | 9 (10) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No